CLINICAL TRIAL: NCT02486484
Title: Phase 2 Ziv-aflibercept in Ocular Disease Short and Long-term Study
Brief Title: Ziv-aflibercept in Ocular Disease Requiring Anti-VEGF Injection
Acronym: Zaltrap
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rafic Hariri University Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Mansour, MD, Clinical Professor, AUB, Chair, Department of Opthalmology, Rafic Hariri Hospital, Rafic Hariri University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RaficHaririUH
Record Dates: First submitted 2015-05-24; First posted 2015-07-01 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Neovascularization; Macular Degeneration; Diabetic Retinopathy; Retinal Vein Occlusion; Choroidal Neovascularization; Retinal Neovascularization; Recurrent Pterygium; Cystoid Macular Edema
Keywords: macular degeneration; diabetic retinopathy; macular edema; retinal vein occlusion; choroidal neovascularization
MeSH Terms: conditions — Neovascularization, Pathologic; Macular Degeneration; Diabetic Retinopathy; Retinal Vein Occlusion; Choroidal Neovascularization; Retinal Neovascularization; Pterygium; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intravitreal ziv-aflibercept (Experimental): intravitreal ziv-aflibercept
  Interventions: Drug: ziv-aflibercept

INTERVENTIONS:
Drug: ziv-aflibercept — zaltrap injection
  Other Names: zaltrap

SUMMARY:
Background/aims: Aflibercept is an approved therapy for neovascular macular degeneration (AMD), diabetic macular edema (DME), retinal vein occlusion and other retinal conditions. Ziv-aflibercept is also approved by FDA and is extremely cost-effective relative to the expensive same molecule aflibercept. In vitro and in vivo studies did not detect toxicity to the retinal pigment epithelium cells using the approved cancer protein, ziv-aflibercept. Ziv-aflibercept had no loss of anti-VEGF activity when kept at 4°C in polycarbonate syringes over 4 weeks. Similar to bevacizumab, compounded ziv-aflibercept would yield a tremendous saving compared to aflibercept or ranibizumab. Phase I studies and case reports did not report any untoward toxic effects but attested to the clinical efficacy of the medication. Our purpose is to ascertain the long-term safety and efficacy in various retinal diseases of intravitreal ziv-aflibercept.

Methods: Prospectively, consecutive patients with retinal disease that require aflibercept (AMD, DME, RVO, and others) will undergo instead the same molecule ziv-aflibercept intravitreal injection of 0.05 ml of fresh filtered ziv-aflibercept (1.25mg). Monitoring of best-corrected visual acuity, intraocular inflammation, cataract progression, and retinal structure by spectral domain OCT to be done initially, one month, 6 months, 1 year, and 2 years after injections.

Anticipated Results: Analyze signs of retinal toxicity, intraocular inflammation, or change in lens status, together with best corrected visual acuity and central foveal thickness at 1 month, 6 months, 1 year and 2 year. Anticipated Conclusions: Off label use of ziv-aflibercept improves visual acuity without ocular toxicity and offers a cheaper alternative to the same molecule aflibercept (or lucentis), especially in the third world similar to bevacizumab.

DETAILED DESCRIPTION:
Ascertain the long term safety and efficacy of ziv-aflibercept in a large variety of ocular diseases and over a long-term after its proven safety and efficacy in the laboratory, in phase one study and in isolated case report.

Background and Significance:

Anti-VEGF therapy is currently one of the mainstay of therapy in a great number of diseases of the eye with intravitreal injections of antiVEGF being the number one procedure done in the office of an ophthalmology practice. The ophthalmic community has currently 2 very expensive antiVEGF both approved by the FDA for ocular use: Ranibizumab and aflibercept. However because of the prohibitive cost of these medications in the third world and the need for repetitive use of these agents in the control of eye disease, the off-label use of bevacizumab is currently the most common anti-VEGF used worldwide because of its equivalent therapeutic efficacy and cost-effective superiority. Bevacizumab and ranibizumab have high affinity to VEGF, aflibercept possess additional properties. Aflibercept (Eylea; Regeneron, Tarrytown, New York, USA and Bayer Healthcare, Leverkusen, Germany) is a fusion protein consisting of the Fc portion of human immunoglobulin IgG1 and the extracellular domains of vascular endothelial growth factor receptors (VEGFR-2 and VEGFR-1), which binds to circulating vascular endothelial growth factor (VEGF), thus acting as a decoy receptor. Laboratory studies and clinical trials suggest that aflibercept's high binding affinity for VEGF may impart greater durability of activity and similar efficacy compared to ranibizumab1 or bevacizumab. Aflibercept is approved by Food and Drug Administration (FDA) for the therapy of wet age related macular degeneration (AMD) , macular edema from retinal vein occlusion or diabetes.3 Ranibizumab is given monthly, while aflibercept is given bimonthly after 3 monthly injections for eyes with wet AMD. Because of the high cost of ranibizumab and aflibercept, a majority of ophthalmologists worldwide tend to treat patients with bevacizumab at a major saving for the patient. Commercially, a much cheaper yet identical fusion protein to aflibercept is ziv-aflibercept. Ziv-aflibercept (Zaltrap, Sanofi-Aventis US, LLC, Bridgewater, NJ and Regeneron Pharmaceuticals, Inc, Tarrytown, NY) was approved by FDA in August 2012 for the treatment of metastatic colorectal carcinoma resistant to an oxiplatin-containing regimen. One may wonder if ziv-aflibercept can be used instead of aflibercept in ophthalmic disorders. Hence the need to answer some major safety concerns: first the difference in osmolarity, and second whether ziv-aflibercept could impair retinal function and alter morphology6. A preliminary study was conducted on the use of ziv-aflibercept in patients with exudative AMD or diabetic macular edema (DME) with poor vision. In addition, the investigators tested the stability of ziv-aflibercept over a period of 4 weeks and the economic implications of the use of compounded drug.

Ziv-aflibercept is supplied in single-use vials of 100 mg per 4 ml and 200 mg per 8 ml formulated as 25 mg/mL ziv-aflibercept in polysorbate 20 (0.1%), sodium chloride (100 mM), sodium citrate (5 mM), sodium phosphate (5 mM), and sucrose (20%), in Water for Injection USP, at a pH of 6.2. Eylea is supplied as a single-use, glass vial designed to deliver 0.05 mL (2mg) of aflibercept (40 mg/mL in 10 mM sodium phosphate, 40 mM sodium chloride, 0.03% polysorbate 20, and 5% sucrose, pH 6.2).

Design and Procedures:

Procedure: inject intravitreal ziv-aflibercept according to published protocols approved by FDA (PROTOCOL A and PROTOCOL B, PROTOCOL C, PROTOCOL D, and other published aflibercept protocols or protocols to be approved or under study for other diseases).

Design: Prospective nonrandomized open label long-term interventional clinical study in patients with subfoveal CNV, extrafoveal CNV due to AMD or other diseases (myopia, inflammatory, angioid streaks, traumatic, idiopathic), DME, BVO or CRVO-related macular edema, diabetic vitreous hemorrhage, and any disease requiring anti-VEGF therapy. The inclusion/exclusion criteria are summarized in tables 1 and 2.

All patients will have to sign a study consent form for the off-label use of intravitreal ziv-aflibercept that is approved by FDA for oncology and the same molecule under different osmolarity for eye disease.

Patients and Methods Patients All patients will have to sign a study consent form for the off-label use of intravitreal ziv-aflibercept.

Pretreatment work up Initial work-up will include best-corrected visual acuity (BCVA) using ETDRS acuity charts, slit-lamp examination of the anterior segment, dilated fundus examination, and fluorescein angiography. Pretreatment macular thickness will be measured with ocular coherence tomography (OCT) for all eyes.

Intravitreal injection of ziv-aflibercept The hospital pharmacy will divide 4cc vial of ziv-aflibercept (ZALTRAP) purchased by the Ophthalmology Department, into twenty 1 cc syringes using aseptic techniques. Therefore, each syringe will contain 0.2 ml of ziv-aflibercept. The syringes will be stored at 4 degrees Celsius for no longer than 30 days. The eye to be treated will be prepared with 5% povidone-iodine solution. Topical Anesthesia will be administered. Using a 30-gauge needle, 0.05 ml ziv-aflibercept will be injected intravitreally through the pars plana 3.5 mm from the limbus. If the intraocular pressure is greater than 25 mmHg or the optic nerve head is not adequately perfused 20 minutes after the injection (if patient reports poor vision of hand motion or less), then a paracentesis will be performed. There is no need to either patch the eye or use topical antibiotics.

Post-injection follow-up Patients will be examined every month after the injection. At each visit, BCVA will be measured along with slit-lamp examination of the anterior segment and dilated fundus examination. OCT will be repeated at each follow-up. The patients will be followed as per the standard approach delineated in the aflibercept trials for AMD or DME. In case of unusually recurrent CNV or DME based on OCT, fluorescein angiography, clinical examination or decrease in vision additional injections may be done depending on the particular case above and beyond the standard protocols. The total follow-up period of the extended study will be 24 months for each patient. Patients and data collection will span over a period of 3 years.

Main outcome The main outcome measures will be improvement in visual acuity, decrease in central retinal thickness, and stability of lesion size in AMD or retinopathy in DME. The paired Student's t-test, Chi-square test, Pearson correlation and ANOVA will be used to analyze the data.

Potential risks Potential risks due to the injection itself are minimal. However patients have about 0.2% risk of eye infection. Retinal detachment and vitreous hemorrhage are extremely rare potential risks. No untoward effects are expected from aflibercept itself. From our experience and others, no signs of ocular toxicity were noted in already treated eyes. But the investigators will again look at any sign of cataract or corneal toxicity. In addition, intraocular inflammation is known to occur at a rate of 0.2% of any anti-VEGF including aflibercept. Such cases will be recorded and treated with anti-inflammatory agents.

PROTOCOL A (AMD) adapted from VIEW 1 and VIEW 2 In eyes with wet AMD, involved eyes are treated every 4 weeks for 3 initial monthly injections, then every 8 weeks till year 1. Patients are evaluated monthly to determine the need for treatment and were treated at least every 12 weeks (capped PRN regimen) 2.

PROTOCOL B (BVO) adapted from VIBRANT The recommended dosage for CRVO is monthly injection till month 6 then monthly monitoring and PRN dosing PROTOCOL C (CRVO) adapted from COPERNICUS and GALILEO The recommended dosage for CRVO is monthly injection till month 6 then monthly monitoring and PRN dosing PROTOCOL D (DME) adapted from VISTA and VIVID The recommended dosage for DME treatment is 5 initial monthly injections followed by one injection every 8 weeks

Subject identification, recruitment, and compensation:

Compensation for participation: None (Compensation relates to 25 times saving of the very expensive drug). The department of ophthalmology would cover the cost of complication from the study, i.e. like treating the patient with endophthalmitis with necessary antibiotics intravitreal and systemic.

Subject identification:

Each collaborator will supply the data with the initials only of the patients to keep patient anonymity under full protection.

Patient recruitment:

Any patient who is a candidate for anti-VEGF therapy for ocular disease is offered this form of therapy such as: choroidal neovascularization of any kind (age-related macular degeneration, myopia, inflammatory, angioid streak, trauma, laser induced, idiopathic) and maculopathy or retinopathy from diabetes mellitus, branch or central retinal vein occlusion, or other occlusive anterior or posterior pole disorders (neovascular glaucoma, rubeosis iridis, corneal neovascularization, angry pterygium, surgical or traumatic fibrovascular ingrowth), and tumor-associated new vessel formation.

Risk/benefit assessment:

There is a risk for endophthalmitis of 0.2% with any intraocular injection. Benefit is visual restoration and avoidance of blindness outweigh the risks

Costs to the subject:

The patient will have a regular charge of the medication (100,000 LL or 66 USD) similar to the off-label use of bevacizumab. Ranibizumab or aflibercept or dexamethasone implants cost each 25 times more, knowing that ziv-aflibercept and aflibercept represent the same molecule exactly. So the investigators are giving the patient the same active product at lower price. This is a major difference between ranibizumab and bevacizumab (different molecule) with 25 times cheaper.

Privacy, Data Storage and Confidentiality:

Confidentiality of the files will be maintained using coded data under the supervision of Dr AMM. Reference between subject code and identity, demographic data, and medical data entered on study sheets will be maintained in a locked drawer in Dr AMM, and on a password-protected computer.

ELIGIBILITY:
Inclusion Criteria: All conditions that require anti-VEGF therapy

1. All eye conditions that require anti-VEGF therapy
2. Ability to understand and sign consent form
3. Ability to come for all follow-ups (2 year followup)
4. Acute form of the disease only in naïve cases

Exclusion Criteria:

1. Cardiovascular, cerebrovascular or peripheral vascular event less than 3 months prior to enrollment
2. Current infection in the eye such as conjunctivitis or keratitis
3. Current upper respiratory tract infection
4. Fever or active body infection
5. Life-threatening disease with short survival
6. late presentation of the disease (chronic end stage disease of the eye)
7. Inability to sign informed consent
8. Inability to come for followups

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
vision before and after ziv-aflibercept | 24 months
  EDTRS

SECONDARY OUTCOMES:
central macular thickness before and after ziv-aflibercept | 24 months
  Optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Mansour, MD, Study Chair — Chair, Department of Ophthalmology, RHUH
Locations (1):
- Rafic Hariri University Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Three-month outcome of ziv-aflibercept for exudative age-related macular degeneration.
  Mansour AM, Chhablani J, Antonios RS, Yogi R, Younis MH, Dakroub R, Chahine H. Br J Ophthalmol. 2016 Mar 30. pii: bjophthalmol-2015-308319. doi: 10.1136/bjophthalmol-2015-308319. [Epub ahead of print] PMID: 27030277

REFERENCES:
- [Background] de Oliveira Dias JR, Xavier CO, Maia A, de Moraes NS, Meyer C, Farah ME, Rodrigues EB. Intravitreal injection of ziv-aflibercept in patient with refractory age-related macular degeneration. Ophthalmic Surg Lasers Imaging Retina. 2015 Jan;46(1):91-4. doi: 10.3928/23258160-20150101-17. PMID 25559518
- [Result] Mansour AM, Al-Ghadban SI, Yunis MH, El-Sabban ME. Ziv-aflibercept in macular disease. Br J Ophthalmol. 2015 Aug;99(8):1055-9. doi: 10.1136/bjophthalmol-2014-306319. Epub 2015 Feb 12. PMID 25677668
- [Result] Mansour AM, Chhablani J, Antonios RS, Yogi R, Younis MH, Dakroub R, Chahine H. Three-month outcome of ziv-aflibercept for exudative age-related macular degeneration. Br J Ophthalmol. 2016 Dec;100(12):1629-1633. doi: 10.1136/bjophthalmol-2015-308319. Epub 2016 Mar 30. PMID 27030277
- [Derived] Mansour AM, Ashraf M, El Jawhari KM, Farah M, Souka A, Sarvaiya C, Singh SR, Banker A, Chhablani J. Intravitreal ziv-aflibercept in diabetic vitreous hemorrhage. Int J Retina Vitreous. 2020 Jan 14;6:2. doi: 10.1186/s40942-019-0204-9. eCollection 2020. PMID 31956432
- [Derived] Mansour AM. Regression of Inflamed Pterygia by Frequent High-Dose Intralesional Ziv-Aflibercept. Cornea. 2017 Aug;36(8):1002-1005. doi: 10.1097/ICO.0000000000001251. PMID 28614154
- See also: ziv-aflibercept in macular disease — http://bjo.bmj.com/cgi/content/full/bjophthalmol-2014-306319